CLINICAL TRIAL: NCT02736149
Title: A Phase 2, Open-Label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Ubenimex in Patients With Pulmonary Arterial Hypertension (WHO Group 1)
Brief Title: Open-Label Extension Study of Ubenimex in Patients With Pulmonary Arterial Hypertension (WHO Group 1)
Acronym: LIBERTY2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following the failure to demonstrate efficacy in EIG-UBX-001, the sponsor decided to terminate Study EIG-UBX-002.
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EIG-UBX-002
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ubenimex

ARMS (1):
- ubenimex (Experimental): ubenimex capsules 150 mg three times a day (TID), administered orally, minimum of 24 weeks for all patients.
  The maximum anticipated time an individual patient will participate will vary because treatment will continue until the last patient enrolled has received at least 24 weeks of open-label treatment.
  Interventions: Drug: ubenimex

INTERVENTIONS:
Drug: ubenimex
  Other Names: UBX

SUMMARY:
Ubenimex is being developed for the treatment of pulmonary arterial hypertension (PAH) (World Health Organization [WHO] Group 1) to improve exercise capacity and delay clinical worsening.

This study is a Phase 2, open-label, extension study to evaluate long-term safety and efficacy of ubenimex in patients with PAH (WHO Group 1) who complete Study EIG-UBX-001.

DETAILED DESCRIPTION:
This study is a Phase 2, open-label, multicenter, extension study to evaluate long-term safety and efficacy of ubenimex in patients with PAH (WHO Group 1) who complete Study EIG-UBX-001 (Study EIG-UBX-001 is a Phase 2, randomized, double-blind, placebo-controlled clinical trial) and meet the eligibility criteria for Study EIG-UBX-002. The primary objective for this study is:

- to obtain long-term safety and tolerability data for ubenimex (150 mg administered three times daily [TID]) in patients with PAH (WHO Group 1).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed Study EIG-UBX-001 through Week 24.
* In the opinion of the Principal Investigator, has been generally compliant with study requirements during Study EIG-UBX-001.
* Agrees to use a medically acceptable method of contraception throughout the entire study period.
* Willing and able to comply with scheduled visits, treatment plans, and laboratory tests and other study procedures.

Exclusion Criteria:

* Is pregnant or lactating.
* Concurrent regular use of another leukotriene pathway inhibitor.
* Any reason that, in the opinion of the investigator, precludes the patient from participating in the study.

  1. Any condition that is unstable or that could jeopardize the safety of the patient and his/her compliance in the study
  2. A serious uncontrolled medical disorder/condition that in the opinion of the investigator would impair the ability of the patient to receive protocol therapy
* An ongoing, drug-related, serious adverse event (SAE).
* Significant/chronic renal insufficiency.
* Transaminases (alanine transaminase, aspartate transaminase) levels >3 × upper limit of normal (ULN) and/or bilirubin level >2 × ULN.
* Absolute neutrophil count <1500 mm3.
* Hemoglobin concentration <9 g/dL at Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (26):
  - California Heart Center Foundation, An Affiliate of Cedars-Sinai Heart Institute, Cedars-Sinai Medical Care Foundation, Beverly Hills, California
  - UCSD Medical Center, La Jolla, California
  - Stanford University Medical Center, Palo Alto, California
  - Harbor - UCLA Medical Center, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - Cleveland Clinic, Florida, Weston, Florida
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Chest Medicine Associates, South Portland, Maine
  - Johns Hopkins University, Pulmonary and Critical Care Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Respiratory Institute, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pennsylvania Medical Center, Pittsburgh, Pennsylvania
  - Alpert Medical School of Brown University Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University Texas Health Science Center, San Antonio, Texas
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario

REFERENCES:
- [Background] Tian W, Jiang X, Tamosiuniene R, Sung YK, Qian J, Dhillon G, Gera L, Farkas L, Rabinovitch M, Zamanian RT, Inayathullah M, Fridlib M, Rajadas J, Peters-Golden M, Voelkel NF, Nicolls MR. Blocking macrophage leukotriene b4 prevents endothelial injury and reverses pulmonary hypertension. Sci Transl Med. 2013 Aug 28;5(200):200ra117. doi: 10.1126/scitranslmed.3006674. PMID 23986401
- [Background] Qian J, Tian W, Jiang X, Tamosiuniene R, Sung YK, Shuffle EM, Tu AB, Valenzuela A, Jiang S, Zamanian RT, Fiorentino DF, Voelkel NF, Peters-Golden M, Stenmark KR, Chung L, Rabinovitch M, Nicolls MR. Leukotriene B4 Activates Pulmonary Artery Adventitial Fibroblasts in Pulmonary Hypertension. Hypertension. 2015 Dec;66(6):1227-1239. doi: 10.1161/HYPERTENSIONAHA.115.06370. Epub 2015 Oct 5. PMID 26558820

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ubenimex
Started | 51
Completed | 0
Not Completed | 51

BASELINE CHARACTERISTICS:
Arm/Group | Ubenimex
Number analyzed (Participants) | 51
Age, Continuous [Mean (Full Range); unit: years] | 51.8 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 46
  More than one race | 0
  Unknown or Not Reported | 3
Mean pulmonary artery pressure [Mean (Standard Deviation); unit: millimetre of mercury (mmHg)] | 45.43 (9.95)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: Number of Patients with TEAEs collected for all patients and recorded on the Adverse Event Case Report Form
Time Frame: At least 24 weeks of open-label treatment with ubenimex followed by 4 weeks follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Ubenimex
Number analyzed (Participants) | 51
Participants | 44

ADVERSE EVENTS:
Time Frame: Up to 24 weeks of treatment from baseline with 4 weeks of follow-up
Groups:
- Ubenimex: ubenimex capsules 150 mg TID, administered orally, minimum of 24 weeks for all patients.
  The maximum anticipated time an individual patient will participate will vary because treatment will continue until the last patient enrolled has received at least 24 weeks of open-label treatment.
Arm/Group | Ubenimex
All-Cause Mortality (participants affected / at risk) | 1/51
Serious Adverse Events (participants affected / at risk) | 12/51
Other Adverse Events (participants affected / at risk) | 42/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ubenimex (N=51)
Right ventricular failure (Cardiac disorders) | 1
Syncope (Vascular disorders) | 1
Device occlusion (General disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Ulcer (General disorders) | 1
Bowel obstruction (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Wound drainage / (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ubenimex (N=51)
Nausea (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
oedema peripheral (Metabolism and nutrition disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6
headache (Nervous system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT02736149/Prot_SAP_000.pdf